CLINICAL TRIAL: NCT07100652
Title: Comparing Different Oxygen Thresholds for Surfactant Administration During Nasal IPPV in Very Preterm Neonates With Respiratory Distress Syndrome: A Superiority RCT
Brief Title: Early Surfactant Administration at FiO₂ >0.25 Under NIPPV for RDS in Very Preterm Infants
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jiulongpo No.1 People's Hospital (Other)
Collaborators: Jiangxi Maternal and Child Health Hospital (Other)
Responsible Party: Principal Investigator, Xingwang Zhu, Jiangxi Maternal and Child Health Hospital, Jiangxi, 337000, China, Jiulongpo No.1 People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Jiangxi Maternal and Child
Record Dates: First submitted 2025-07-27; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Respiratory Distress Syndrome (&Amp; [Hyaline Membrane Disease])
MeSH Terms: conditions — Respiratory Distress Syndrome; Hyaline Membrane Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lower oxygen threshold group (FiO₂ >0.25) (Experimental): Surfactant was administered as a single initial dose when the fraction of inspired oxygen (FiO₂) exceeded 0.25
  Interventions: Procedure: Threshold FiO₂
- Higer oxygen threshold group (FiO₂ >0.3) (Active Comparator): Surfactant was administered as a single initial dose when the fraction of inspired oxygen (FiO₂) exceeded 0.3
  Interventions: Procedure: Threshold FiO₂

INTERVENTIONS:
Procedure: Threshold FiO₂ — Group 1 (Intervention Group) received the initial dose of pulmonary surfactant immediately upon reaching an inhaled oxygen concentration (FiO₂) >0.25.
  Group 2 (Control Group) received the initial dose of pulmonary surfactant as early as possible within 48 hours, but only when FiO₂ was titrated to >0.3 based on the infant's clinical condition.

SUMMARY:
This multicenter randomized controlled trial investigates whether initiating pulmonary surfactant (PS) at a lower oxygen threshold (FiO₂ >0.25) during nasal intermittent positive pressure ventilation (NIPPV) for very preterm infants with respiratory distress syndrome (RDS) reduces noninvasive ventilation failure rates (primary outcome: intubation requirement), compared to the standard threshold (FiO₂ >0.3). By establishing the clinical superiority of early PS administration, this study aims to refine evidence-based guidelines for RDS management in preterm neonates.

ELIGIBILITY:
Inclusion Criteria:

* (1) Gestational Age: 26 weeks +0 day to 31 weeks+6days at birth (inclusive). (2) Clinical Diagnosis of NRDS: Symptoms: Tachypnea, grunting, and/or progressive respiratory distress. Imaging Findings: Chest X-ray showing at least one of: Ground-glass opacity, Air bronchograms, Diffuse "white lung" pattern, Lung Ultrasound (recommended).

  (3) Admission to NICU within 3 hours of birth. Requirement for non-invasive nasal intermittent positive pressure ventilation (NIPPV) at enrollment.

  (4) Signed informed consent obtained from parent(s) or legal guardian(s).

Exclusion Criteria:

1. Invasive mechanical ventilation during delivery or transport to NICU.
2. Structural upper airway abnormalities precluding non-invasive ventilation.
3. Confirmed diagnosis of major congenital malformations
4. Endotracheal intubation for indications unrelated to NRDS (e.g., surgery, sepsis management)
5. Initiation of non-invasive ventilation >3 hours post-birth.
6. Voluntary discharge or treatment withdrawal within 72 hours post-enrollment.
7. Parental/guardian refusal to Sign informed consent or Authorize surfactant administration
8. Incomplete clinical records or missing key outcome variables

   -

Max Age: 3 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 384 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Non-invasive respiratory support failure, defined by the need for IMV within 72 after birth | 72 hours after birth

SECONDARY OUTCOMES:
The requirement for repeated pulmonary surfactant administration, including the total number of doses utilized | 7 days after birth
BPD, defined according to the NICHD definition | 3 months after birth
airleaks occurred after the extubation | 3 months after birth
retinopathy of prematurity (ROP) > 2nd stage | 3 months after birth
necrotizing enterocolitis (NEC) ≥ 2nd stage | 3 months after birth
IVH > 2nd grade | 3 mionths after birth
hemodynamically significant patent ductus arteriosus (PDA) | 3 months after birth
weekly weight gain (in grams/d) for the first 4 weeks of life or until NICU discharge, whichever comes first. | 3 months after birth
Duration of non-invasive respiratory support | 3 months after birth
total hospitalization cost | 6 months after birth
nasal skin injury | 3 months after birth
in-hospital mortality | 6 months after birth
ventilator-free days | 3 months after birth

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangxi Maternal and Child Health Hospital, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Derived] Yang R, Fang Z, Liu KZ, Zhu X, Ding XP, Luo Q, Zhou WJ, Hu XW, Zhou JL, Tang WY, Shi Y. Comparison of two fractions of inspired oxygen thresholds (0.25 vs 0.30) for surfactant administration in very preterm infants with respiratory distress syndrome under nasal intermittent positive pressure ventilation: study protocol for a multicentre randomised controlled, superiority trial. BMJ Paediatr Open. 2025 Nov 10;9(1):e003998. doi: 10.1136/bmjpo-2025-003998. PMID 41213831